CLINICAL TRIAL: NCT06115512
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of a Single Lntervertebral Local Administration of AGA111 in Patients With Degenerative Disc Disease Undergoing Lumbar Lnterbody Fusion
Brief Title: A Phase 3 Study of AGA111 in Patients With Degenerative Disc Disease Undergoing Lumbar Interbody Fusion
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Angitia Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT22-001
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGA111 (Experimental): AGA111 in autologous blood coagulum (ABC) is locally delivered at the intervertebral space.
  Interventions: Drug: AGA111
- Placebo (Placebo Comparator): Placebo in ABC is locally delivered at the intervertebral space.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGA111 — AGA111 is locally administered in an ABC carrier at the intervertebral space during the lumbar interbody fusion.
  Arms: AGA111
Drug: Placebo — Placebo is locally administered in an ABC carrier at the intervertebral space during the lumbar interbody fusion.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the overall efficacy of a single intervertebral local administration of AGA111 in patients with degenerative disc disease undergoing lumbar interbody fusion.

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of a single intervertebral local administration of AGA111 in patients with degenerative disc disease undergoing lumbar interbody fusion. About 400 subjects who meet the eligibility criteria will be randomly assigned to the following two treatment groups in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease of L3-S1 with low back pain, with or without a history of radiating leg or buttock pain, paresthesia, numbness or weakness secondary to radiculopathy of the corresponding spinal segment;
2. Has radiographic evidence (e.g., X-ray and CT/magnetic resonance imaging MRI) of degenerative disc disease;
3. Adults ≥ 18 and ≤ 80 years of age and skeletally mature at the time of surgery;
4. Plan to undergo a single-level lumbar interbody fusion;
5. Preoperative ODI score ≥ 30;
6. Has not respond to conservative treatment (e.g, bed rest, physical therapy, drugs, local injections, manipulation and other non-surgical treatments) for a period of at least 3 months;
7. Willing and able to comply with the protocol and able to understand and sign the subject's informed consent form (ICF) ;
8. Female subjects of child-bearing potential must agree to use a highly effective method of birth control during the study and for 1 year after the administration of investigational drug, and must have a negative pregnancy test prior to the randomization.

Exclusion Criteria:

1. Has undergone other decompression, fusion, and/or other non-fusion spinal surgery at the spinal segment intended to undergo the surgery prior to the screening (except for transforaminal endoscopic discectomy);
2. Known other significant lumbar instability;
3. Lumbar scoliosis > 30 degrees (evaluated by investigators);
4. Presence of active malignancy or prior history of malignancy;
5. Overt or active infection, either local to surgical space or systemic;
6. Patients with a dual-energy X-ray absorption (DXA) total hip T-score ≤ -3.0;
7. Body weight index (BMI) <18.5 kg/m2 or BMI > 35 kg/m2;
8. Have received other treatments affecting fusion surgery, such as radiotherapy near the surgical site;
9. Presence of other co-morbidities of the spine or upper/lower extremities that may affect the investigator's assessment of the lumbosacral nervous system and/or pain;
10. Presence of mental disease or psychiatric condition that interferes with the patient's self-assessment of function, pain, or quality of life;
11. History of progressive osseous heteroplasia or fibrodysplasia ossificans progressiva;
12. Known hypersensitivity or allergy to bone morphogenetic protein (BMP) products or their excipient; and/or instrumentation materials in surgery, e.g., titanium, titanium alloy, cobalt chrome, cobalt chrome alloy, or polyetheretherketone (PEEK);
13. Pregnant or lactating women; or plan to become pregnant within 1 year following the study surgery.
14. Other conditions that, in the opinion of the investigator, would interfere with the subject's ability to comply with the protocol, and other conditions that will make the subject inappropriate for participation in the study as judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall success rate: Proportion of subjects who achieve overall success. | Up to 52 weeks

SECONDARY OUTCOMES:
Success rate of radiographic fusion | Up to 52 weeks
Mean change of ODI (Oswestry Disability Index) score | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angitia Medical Director, Study Director — Angitia Biopharmaceutics Guangzhou Limited
Locations (35):
- China (35):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - Zhejiang Provincial People's Hospital Bijie Hospital, Bijie, Guizhou
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Tongji Hospital, Tongji Medical College, Huazhong Universit of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shenyang Orthopedics Hospital, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Xi'an Honghui Hospital, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No